CLINICAL TRIAL: NCT06988969
Title: Factors Influencing Vaccine Hesitancy Among Parents of Children Aged 0-48 Months: A Machine Learning Prediction
Brief Title: Predicting Vaccine Hesitancy Using Machine Learning
Status: Active, not recruiting | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Emel AVÇİN, Ass Prof, University of Yalova
Other Study IDs: Emel Avcin MLT
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Vaccine Refusal; Vaccine Hesitancy; Machine Learning; Children
Keywords: Children; Vaccines; Hesitancy; Machine learning; Immunization; Parent
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents of children aged 0-48 months: Parents who meet the following criteria will be included in the study: those who have proficiency in understanding and reading the Turkish language; are 18 years of age or older; have children aged 0-4 years; are able to use technological devices such as mobile phones or computers to access social media platforms (Participants used social media platforms such as Instagram and WhatsApp to communicate) via the internet; consent to participate in the study; and whose children do not have any absolute contraindications for vaccination.

SUMMARY:
In recent years, emerging technologies such as the Internet of Things (IoT), Artificial Intelligence (AI), and Virtual Reality (VR) have rapidly become integrated into daily life. The widespread use of these applications has led to the accumulation of vast amounts of data, giving rise to what is commonly referred to as "Big Data." Due to the sheer volume, manual processing and analysis of these large datasets are not feasible. Therefore, software tools and libraries-such as Python and R libraries-have been developed to perform these analyses efficiently and to generate predictions for the future by leveraging historical data through Machine Learning (ML) algorithms.

The primary goal of machine learning algorithms is to discover patterns within existing data and use these patterns to make accurate predictions on new data. The use of machine learning in the field of healthcare has gained significant momentum in recent years. However, a review of the literature reveals that research specifically addressing childhood vaccine hesitancy remains limited.

This study aims to identify the factors contributing to vaccine hesitancy among parents of children aged 0-48 months and to develop a predictive model using machine learning techniques based on these factors. Such a model could help anticipate the likelihood of vaccine refusal among parents and thereby support the development of targeted public health strategies for at-risk populations.

ELIGIBILITY:
Inclusion Criteria:

Parents who meet the following criteria will be included in the study:

* Have proficiency in understanding and reading the Turkish language,
* Are able to use technological devices such as mobile phones or computers to access social media platforms (Participants used social media platforms such as Instagram and WhatsApp to communicate) via the internet,
* Are 18 years of age or older,
* Have children aged 0-4 years,
* Consent to participate in the study,
* Have children without any absolute contraindications to vaccination.

Exclusion Criteria:

* Parents of high-risk infants (such as those with a history of systemic illness, preterm labor, anomalies, etc.),
* Parents who are unwilling to participate in the study will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No sample size calculation was performed in this study. Between June 2025 and September 2025, all parents of children aged 0-4 years who met the inclusion criteria and could be reached with the questionnaires were included in the study. Snowball sampling method will be used to reach the parents. The study population consists of parents who have children aged 0-4 years, possess proficiency in understanding and reading the Turkish language, and can be accessed via social media platforms using technological devices.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Parental Vaccine Hesitancy Status | Day 1 (Parents will be sent the questionnaire and asked to respond promptly.)
  The Vaccine Hesitancy Scale is a measurement tool designed to assess individuals' vaccine hesitancy or opposition. It consists of 21 items across 4 subscales and uses a 5-point Likert scale format. The four subscales of the scale are: Vaccine Benefit and Protective Value, Vaccine Opposition, Solutions for Avoiding Vaccination, and Justification of Vaccine Hesitancy. Higher scores on the scale indicate greater levels of vaccine hesitancy or opposition.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL AVÇİN, Assist Prof, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)